CLINICAL TRIAL: NCT06420232
Title: Protocol for Using a Weighted Blanket to Treat Anxiety Related to Trying New Foods in the Pediatric Population
Brief Title: Weighted Blanket to Treat Anxiety Related to Trying New Foods the Pediatric Population
Acronym: Food Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: challenges with recruitment and attrition, and PI graduated from UTMB PPOTD program
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0342
Record Dates: First submitted 2024-05-10; First posted 2024-05-17 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Food Neophobia; Picky Eating; Avoidant Restrictive Food Intake Disorder; Anxiety State
Keywords: weighted blanket; food avoidance; picky eater; state anxiety; anxiety related to food; children
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Food Fussiness; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: usual care waitlist control period followed by one month intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Weighted Blanket (Experimental)
  Interventions: Device: weighted blanket

INTERVENTIONS:
Device: weighted blanket — Blanket weighted with 10% or less of body weight applied to child prior to meals for duration no more than 15 minutes

SUMMARY:
This small experimental pilot study addresses the knowledge gap related to the use of weighted blankets for children with anxiety related to food and eating.

DETAILED DESCRIPTION:
The purpose of the study is to research if weighted blankets might help children with anxiety related to food tolerate new foods better. The parent will be asked to complete a 10-question questionnaire and make a list of the foods the child eats on three occasions (before the study begins, after a control period and after the child uses the weighted blanket). The child will be asked to use a weighted blanket for 5 to 15 minutes prior to at least 3 meals a week for one month, and the child will be asked to complete a 20-question questionnaire taking about 5-12 minutes to complete asking about how they feel on days that they use the weighted blanket and one time a week during the month that they don't use the weighted blanket. The parent will be asked to report any new foods the child tries on the days that they do use the weighted blanket. The parent will be asked to keep the weighted blanket and supervise all use of the weighted blanket for safety. This study will take approximately 2 months total.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and guardian has provided informed consent in a manner approved by the IRB and is willing and able to comply with the trial procedures.
2. Subject has identified feeding challenges
3. Subject has anxiety related to food as reported by caregiver
4. Subject is between the ages of 8-12
5. Subject has good reading abilities
6. Subject weighs 30 pounds or more

Exclusion Criteria:

1. Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation due to the inability to remove the blanket safely. Examples of diagnoses that would exclude a participant include spinal cord injury, cerebral palsy, and muscular dystrophy.
2. Concurrent participation on another research study
3. Participants outside of the ages 8-12
4. Participants refuse to use the weighted blanket
5. If the use of a weighted blanket is contraindicated for any reason
6. Participants lacking the reading ability to complete a questionnaire
7. Participants who weigh under 30 pounds per parent report and cannot use a commercially available weighted blanket as the minimum weight of a weighted blanket is 3 pounds will be excluded but this exclusion is unlikely due to the inclusion age range

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Area Speech & Occupational Therapy, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
upon request, deidentified data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: May 2025 for 5 years
Access Criteria: per request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weighted Blanket
Started | 6
Control Period (The control period consists of usual care occupational therapy services lasting 1 month prior to the treatment period.) | 6
Treatment Period (The treatment period consists of usual care occupational therapy services and weighted blanket use lasting 1 month after the control period.) | 3
Completed | 3
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Weighted Blanket
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Food Neophobia Scale for Children Questionnaire
Description: The Food Neophobia Scale for Children is a 10-item Likert scale questionnaire that parents complete. The responses to the questions on the Food Neophobia Scale for Children ranged from one (Strongly Agree) to seven (Strongly Disagree). The value of each response could be worth 7 points, depending on the responses. The caregivers completed the Food Neophobia Scale for Children questionnaire at baseline, following the usual care period, and after the intervention period. Higher total scores indicate higher levels of food neophobia. The total score range was 10 (lowest) to 70 (highest).
Time Frame: Baseline, prior to treatment and post treatment
Population: One participant did not complete the FNSC questionnaire at post-treatment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Weighted Blanket
Number analyzed (Participants) | 2
score on a scale
  Baseline | 67.5 (2.12132)
  Prior Treatment without the blanket | 67 (1.414214)
  Post Treatment with the blanket | 65 (1.414214)

2. Primary Outcome: State-Trait Anxiety Inventory for Children (STAIC) Median T-Score
Description: The STAI-C Anxiety Scale asks for ratings of agreement on a 3-point scale using the stem "I feel…" for 20 items both indicative of the presence of anxiety (e.g., 1= not upset; 2= upset; 3= very upset) and reverse-worded (e.g., 1= very calm; 2= calm; 3= not calm) items. The participants completed the STAIC S-Anxiety scale three times per week during the usual care and treatment period. Higher T-scores indicate higher anxiety. The mean of the normalized T-score was 50, and the standard deviation was 10. No established clinical thresholds are defined for this measure.
Time Frame: Prior and post treatment, up to 2 months
Measure: Median (Standard Error); unit: T-score
Arm/Group | Weighted Blanket
Number analyzed (Participants) | 3
T-score
  Prior to Treatment | 57 (34.69577)
  Post Treatment | 54.5 (34.63697)

3. Primary Outcome: Average Number of New Foods
Description: The average number of foods tried during the control period will be compared to baseline and the average number of new foods tried during the control period will be compared to the average number of new foods tried in the treatment period to understand if more foods were tried when using the weighted blanket.
Time Frame: Control Period (1 month) and Treatment Period (1 month)
Measure: Mean (Standard Error); unit: number of foods tried
Arm/Group | Weighted Blanket
Number analyzed (Participants) | 3
number of foods tried
  Control Period | 7 (2.645751)
  Treatment Period | 6 (2)

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Treatment Period: A blanket weighted with 10% or less of body weight is applied to a child prior to meals for a duration of no more than 15 minutes 3 times a week for a period of 1 month.
- Control Period: Occupational therapy services treatment as usual without use of a weighted blanket for a period of 1 month.
Arm/Group | Treatment Period | Control Period
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Challenges with recruitment and attrition, and PI graduated from the UTMB PPOTD program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT06420232/Prot_SAP_000.pdf